CLINICAL TRIAL: NCT00440609
Title: A Phase I/II Study Comparing the Treatment of Clinically Significant Diabetic Macular Edema (CSDME) With 0.5mg Ranibizumab, 1.0mg Ranibizumab and 2.0mg Ranibizumab
Brief Title: Study Comparing 0.5mg of Ranibizumab and Higher Doses in the Treatment of Clinically Significant Diabetic Macular Edema
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Philip J. ferrone, M.D. (Other)
Responsible Party: Sponsor-Investigator, Philip J. ferrone, M.D., Prinicpal Investigator, Long Island Vitreoretinal Consultants
Organization: Long Island Vitreoretinal Consultants (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FVF3802s
Record Dates: First submitted 2007-02-23; First posted 2007-02-27 (Estimated); Last update posted 2013-08-02 (Estimated); Status verified 2013-08

CONDITIONS: Clinically Significant Diabetic Macular Edema
MeSH Terms: interventions — Ranibizumab

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 0.5mg transitioning to 2.0mg (Active Comparator): Ranibizumab-intravitreal injection
  Interventions: Drug: ranibizumab
- 1.0 mg transitioning to 2.0mg (Active Comparator): Ranibizumab-intravitreal injection
  Interventions: Drug: ranibizumab

INTERVENTIONS:
Drug: ranibizumab — 0.5mg or 1.0mg intravitreal injection given monthly for 3 months then every other month if needed, for the first year.Patients may be treated monthly as needed. Patients in Cohort 1(the first 30 patients)will be eligible to receive treatment as needed with 2.0mg ranibizumab starting at month 24. Patients in Cohort 2(the remaining 20)will be eligible to receive treatment as needed with 2.0mg ranibizumab starting at month 12.Patients may receive 2.0mg ranibizumab for a period limited to 24 months following administration of the first 2.0mg dose. Patients completing 36 months will be eligible to be followed for an additional 24 months. Starting at Month 36, patients will be able to receive monthly, the assigned dose that they received/or could have received(if re-treatment criteria was met)at Month 35. 2/1/12 - the 2.0mg dose has been discontinued, all subjects will transition to the 0.5mg dose.

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of Ranibizumab in patients with Clinically Significant Diabetic Macular Edema (CSDME). It will also compare treatment outcomes for patients receiving 0.5mg Ranibizumab and higher doses of 1.0mg and 2.0mg Ranibizumab.

ELIGIBILITY:
Inclusion Criteria:

* Type I or Type II diabetic subjects
* Vision between 20/20 and 20/400
* Presence of Clinically Significant Diabetic Macular Edema

Exclusion Criteria:

* Presence of any condition that would prevent clear visualization of the back of the eye
* Uncontrolled glaucoma
* Complications of glaucoma
* Inflammation inside the eye
* Certain prior eye surgeries, other than cataract surgery
* Other eye diseases that may compromise the vision in the study eye
* Certain prior eye treatments
* Pregnancy
* Uncontrolled health conditions
* History of heart attack
* History of stroke
* Current participation in another investigational trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2007-03; Primary Completion 2012-11 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
To evaluate safety and tolerability of ranibizumab in patients with clinically significant diabetic macular edema | month 12
To compare the treatment of clinically significant diabetic macular edema with 0.5 mg of ranibizumab to 1.0 mg ranibizumab | month 12

SECONDARY OUTCOMES:
Mean change in visual acuity as measured by ETDRS from baseline to month 12, 24 36,48 and 60 in each arm. | month 12, 24, 36, 48 and 60
Mean change in central retinal thickness on OCT from baseline to month 12, 24, 36, 48 and 60 in each arm | month 12, 24, 36,48 and 60
Changes observed on the fluorescein angiogram in each arm | Month 60
Mean number of ranibizumab injections required in each arm | Month 60
The need for "rescue therapy" with laser in each arm | Month 60
Evaluate the efficacy and safety of ranibizumab in the fellow eye in the sub-group of patients who require treatment for clinically significant diabetic macular edema in the fellow eye | Month 60

CONTACTS AND LOCATIONS:
Overall Officials: Philip J. Ferrone, MD, Principal Investigator — Long Island Vitreoretinal Consultants
Locations (2):
- United States (2):
  - Long Island Vitreoretinal Consultants, Great Neck, New York
  - Long Island Vitreoretinal Consultants, Hauppauge, New York